CLINICAL TRIAL: NCT03845036
Title: The Effects of Diet and Exercise Interventions in Peripheral Artery Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Milton S. Hershey Medical Center (Other); National Institute on Aging (NIA) (NIH); Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16383; R01AG070086-01A1 (NIH)
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Claudication; Peripheral Artery Disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DASH Diet plus Home-Based Exercise (Experimental): The DASH dietary program consists of a diet emphasizing foods rich in fruits, vegetables, whole grains, and low-fat dairy, in which patients record daily servings of fruits and vegetables. The home-based exercise program consists of intermittent walking to moderate claudication pain 3 times per week for 3 months in a home-based setting.
  Interventions: Behavioral: DASH Diet plus Home-Based Exercise
- Home-Based Exercise (Active Comparator): The home-based exercise program consists of intermittent walking to moderate claudication pain 3 times per week for 3 months in a home-based setting.
  Interventions: Behavioral: Home-Based Exercise

INTERVENTIONS:
Behavioral: DASH Diet plus Home-Based Exercise — The DASH dietary program consists of a diet emphasizing foods rich in fruits, vegetables, whole grains, and low-fat dairy, in which patients record daily servings of fruits and vegetables. The home-based exercise program consists of intermittent walking to moderate claudication pain 3 times per week for 3 months in a home-based setting.
  Arms: DASH Diet plus Home-Based Exercise
Behavioral: Home-Based Exercise — The home-based exercise program consists of intermittent walking to moderate claudication pain 3 times per week for 3 months in a home-based setting.
  Arms: Home-Based Exercise

SUMMARY:
This study is a 3-month, prospective, randomized controlled clinical trial designed to address the efficacy of the DASH dietary program combined with a home-based exercise program, quantified by a step activity monitor, to improve exercise and vascular outcome measures in patients with PAD.

DETAILED DESCRIPTION:
This study seeks to (1) compare the changes in 6-minute walk distance (6MWD) and physical function quality of life in patients with peripheral artery disease (PAD) following a combined intervention of the dietary approaches to stop hypertension (DASH) dietary program plus a home-based exercise program, and following a home-based exercise program alone; and (2) compare the changes in microvascular function and inflammation in patients following the combined DASH diet and home-based exercise program, and the home-based exercise program alone.

The investigators hypothesize that the combined DASH diet and exercise program will result in greater increases in 6MWD and in the physical function quality of life than the exercise program alone. Further, it is hypothesized that the combined DASH diet and exercise program will result in greater improvements in calf muscle oxygen saturation [StO2] following exercise, and in high-sensitivity C-reactive protein (hsCRP]) than the exercise program alone.

The home-based exercise program consists of intermittent walking to moderate claudication pain in a home-based setting. The DASH dietary program consists of the dietary approaches to stop hypertension diet emphasizing foods rich in fruits, vegetables, whole grains, and low-fat dairy.

ELIGIBILITY:
Inclusion Criteria:

1. History of claudication,
2. Presence of PAD, defined by meeting at least one of the following criteria (ABI at rest < 0.90, or > 20% decrease in ABI following a heel-rise exercise test in patients with a normal ABI at rest (> 0.90), or history of peripheral revascularization.

Exclusion Criteria:

1. absence of PAD, defined by meeting all of the following 3 criteria (ABI at rest > 0.90), < 20% decrease in ABI following a heel-rise exercise test, and no history of peripheral revascularization,
2. non-compressible vessels (ABI > 1.40),
3. rest pain due to PAD (Fontaine stage III; Rutherford Grade II),
4. tissue loss due to PAD (Fontaine stage IV; Rutherford Grade III),
5. use of medications indicated for the treatment of intermittent claudication (cilostazol and pentoxifylline) initiated within three months prior to investigation,
6. peripheral revascularization within one month prior to investigation,
7. active cancer,
8. end stage renal disease defined as stage 5 chronic kidney disease,
9. medical conditions that are contraindicative for exercise according to the American College of Sports Medicine,
10. cognitive dysfunction (mini-mental state examination score < 24), and
11. failure to complete the baseline tests within three weeks.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Peak Walking Time | 3 months
  The change in the time walked on a treadmill test
Physical Function subscale of quality of life from the Medical Outcomes Study Short-Form 36 questionnaire | 3 months
  The change in the Physical Function subscale from the pre-test value to the post-test value

SECONDARY OUTCOMES:
calf muscle oxygen saturation | 3 months
  The change in the calf muscle oxygen saturation value during exercise from the pre-test value to the post-test value
6-minute walk distance | 3 months
  The change in 6-minute walk distance from the pre-test value to the post-test value
high-sensitivity C-reactive protein | 3 months
  The change in the high-sensitivity C-reactive protein value from the pre-test value to the post-test value

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Gardner, Ph.D., Principal Investigator — Professor, Department of Medicine, Cardiology
Locations (1):
- O'Donoghue Research Building, University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gardner AW, Parker DE, Montgomery PS, Scott KJ, Blevins SM. Efficacy of quantified home-based exercise and supervised exercise in patients with intermittent claudication: a randomized controlled trial. Circulation. 2011 Feb 8;123(5):491-8. doi: 10.1161/CIRCULATIONAHA.110.963066. Epub 2011 Jan 24. PMID 21262997
- [Result] Gardner AW, Parker DE, Montgomery PS, Blevins SM. Step-monitored home exercise improves ambulation, vascular function, and inflammation in symptomatic patients with peripheral artery disease: a randomized controlled trial. J Am Heart Assoc. 2014 Sep 18;3(5):e001107. doi: 10.1161/JAHA.114.001107. PMID 25237048
- [Result] Gardner AW, Bright BC, Ort KA, Montgomery PS. Dietary intake of participants with peripheral artery disease and claudication. Angiology. 2011 Apr;62(3):270-5. doi: 10.1177/0003319710384395. PMID 21406424